CLINICAL TRIAL: NCT02884752
Title: Retrospective Study of Bone Infection Due to Campylobacter Spp
Acronym: CAMPYLO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Centre de Référence des Infections Ostéo-Articulaires du Grand Ouest (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAMPYLO
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Campylobacter Infections; Bone Diseases, Infectious
MeSH Terms: conditions — Campylobacter Infections; Bone Diseases, Infectious

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Only 24 cases of Campylobacter bone and joint infection (BJI) have been reported worldwide between 1955 and 2008. Between 2010 and 2012, 7 cases were observed in two University hospitals in France. This increasing number of cases raises several issues. Are they the consequences of better detections and reporting, or are they reflecting any epidemiologic changes? For answering these questions, we performed a 10 year (2002-2012) retrospective multicenter (6 centers) study on BJI (native and implanted joints) due to Campylobacter species.

DETAILED DESCRIPTION:
Methods: By browsing the microbiological database of 6 BJI French reference centers, we collected all cases due to Campylobacter species between 2002 and 2012, including first and relapse cases. Clinical, microbiological and treatment features were analyzed using descriptive statistics.

Results: 14 episodes of BJI due to Campylobacter spp were identified in 10 patients. Mean age was 76.8 y.o. (63-96). Sex ratio M/F was 1.5. Nine patient had hip (n=6), knee (n=2), and shoulder (n=2) implants. Immunosuppression was observed in 6 patients (3 cancers, 1 cirrhosis, 1 rheumatoid arthritis, 1 corticosteroid treatment). During the 10 primary cases: all patients had fever and 2 presented digestive symptoms. Campylobacter spp were isolated on per operative samples in 5 patients. One of them presented positive blood culture. 5 patients had joint punctures: all of them were positives. Campylobacter species were C. fetus (n=7), C. coli (n=2) and C. spp (1). Strains were resistant to nalidixic acid (=10), ciprofloxacin (n=4), erythromycin (n=3) or cefotaxime (n=2). Only one C. fetus was susceptible to all antibiotics tested. Surgical treatment was performed in 8 patients (2 two-stage procedure, 6 irrigation). The mean duration of adapted antibiotherapy was 77 days (26-237). 3 out of 4 relapse cases were due to C. fetus. All were resistant to more than one antibiotic classes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with peroperative bone samples positive to Campylobacter spp. between Jan 2002 and Dec. 2012
* Adults over 18 yo
* No opposition to the study expressed by the patient

Exclusion Criteria:

* Adults below 18 yo
* Spine infection to Campylobacter spp.
* Outside of the timeframe of the study
* No microbiologic data available
* Opposition to the study expressed by the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with peroperative bone samples positive to Campylobacter spp.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate of reported prosthetic joint Campylobacter spp. Infections | 1986 to 2013

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Ansart, MD, PHD, Principal Investigator — CHU Brest
Locations (1):
- CHRU de Brest, Brest, France